CLINICAL TRIAL: NCT02056379
Title: Comparison Between Inhaled Budesonide and Intravenous Dexamethasone Treatments for Postextubation Stridor in Children
Brief Title: Comparison Between Budesonide and Dexamethasone Treatments for Respiratory Discomfort After Extubation on Children
Acronym: BUDEXA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Hospital M'Boi Mirim (Other)
Responsible Party: Principal Investigator, Daniela Nasu Monteiro Medeiros, MD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 508177
Record Dates: First submitted 2014-01-23; First posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Stridor
Keywords: stridor; laryngitis; budesonide; dexamethasone; children
MeSH Terms: conditions — Respiratory Sounds; Laryngitis | interventions — Budesonide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide (Active Comparator): 2 mg of nebulized budesonide at 12/12 hours and 8 cc of intravenous normal saline.
  Interventions: Drug: Budesonide
- Dexamethasone (Active Comparator): This group will receive 0,15 mg/kg/dose of intravenous dexamethasone at 6/6 hours and 8 cc of nebulized normal saline at 12/12 hours.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Budesonide — The subjects will receive a 5 ml normal saline inhalation right after extubation and will be re-evaluated in 5 to 10 minutes. The ones who develop upper airway obstruction and stridor with a Downes-Raphaelly score of 2 or higher will receive 0.5 ml/kg of inhaled epinephrine 1:1000 diluted to a final volume of 5 ml with a maximum dose of 2.5 ml in children up to 4 years and 5 ml in children with 5 years and above, as recommended by the American Academy of Pediatrics. The subjects who do not show an improvement after the epinephrine treatment will then be randomized to receive 2 mg of inhaled budesonide and 3 ml of IV normal saline. If there is an improvement the following maintenance therapy will be instituted for 48 hs and the subjects will receive 2 mg of budesonide q12hs and 3 ml of IV NS q6hs.
  Other Names: Pulmicort
  Arms: Budesonide
Drug: Dexamethasone — The subjects will receive a 5 ml normal saline inhalation right after extubation and will be re-evaluated in 5 to 10 minutes. The ones who develop upper airway obstruction and stridor with a Downes-Raphaelly score of 2 or higher will receive 0.5 ml/kg of inhaled epinephrine 1:1000 diluted to a final volume of 5 ml with a maximum dose of 2.5 ml in children up to 4 years and 5 ml in children with 5 years and above, as recommended by the American Academy of Pediatrics. The subjects who do not show an improvement after the epinephrine treatment will then be randomized to receive 8 ml of inhaled normal saline and 0.6 mg/kg of IV dexamethasone. The dexamethasone group will receive 8 ml of inhaled NS q12hs and 0.15 mg/kg/dose of dexamethasone q6hs.
  Other Names: Decadron, Hexadrol, Maxidex
  Arms: Dexamethasone

SUMMARY:
The study aims to analyze and compare the clinical effects of using inhaled budesonide or intravenous dexamethasone in the treatment of postextubation stridor on children admitted to the pediatric intensive care units at Hospital Municipal do M´Boi Mirim and Hospital Albert Einstein.

DETAILED DESCRIPTION:
The investigators propose to perform a prospective, randomized, controlled and double-blind non inferiority study enrolling 70 children with postextubation stridor. The population will be divided in two groups: group 1 will receive inhaled budesonide and IV NS (intravenous normal saline) and group 2 will receive IV (intravenous) dexamethasone and inhaled normal saline. The study aims to analyze and compare (I would just say compare) the clinical effects of using inhaled budesonide or IV dexamethasone in the treatment of postextubation stridor on children admitted to the pediatric intensive care units at Hospital Municipal do M´Boi Mirim and Hospital Albert Einstein.

ELIGIBILITY:
Inclusion Criteria:

* patients intubated for periods longer than 24hs
* age between 28 days and than 15 years
* post extubation stridor must be clinically diagnosticated by a MD
* informed consent must be obtained

Exclusion Criteria:

* patients under palliative care
* presence of neuromuscular disease
* previous airway pathologies
* epiglottitis, aspiration of foreign bodies
* viral laryngitis
* former airway surgery
* patients previously included in the study within the same hospital admission
* corticosteroid use in the 48hs preceding extubation

Ages: 1 Month to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The decrease of stridor and respiratory discomfort | 6 hours
  The investigators will use the Downes-Raphaelly score as an objective measurement tool of degree of respiratory discomfort. The decrease of Downes-Raphaelly score will be considered as an improvement of patient condition.

SECONDARY OUTCOMES:
Number of patients with adverse events | 1 day
  The investigators will consider hypertension, hyperglycemia, gastrointestinal hemorrhage as adverse events of the usage of dexamethasone.
The time frame of stridor's and respiratory discomfort's improvements | 1 hour
  The investigators will study if budesonide has the same time frame improvement treating stridor and respiratory discomfort.
The number of patients that will have extubation failure at each arm | 2 days
  Extubation failure will be considered as a need for re-intubation during de 48 hours after extubation.
The number of inhaled epinephrine doses used in each arms. | 2 days
  The inhaled epinephrine will be used as rescue therapy to absence of improvement. The number of inhaled epinephrine dosage used on each patient will be a measure of efficacy of budesonide or dexamethasone.
The number of patients who need for non invasive mechanical ventilation or Heliox | 2 days
  The non invasive mechanical ventilation and Heliox are rescue therapies. The number of patients treated with those rescue therapies will be a measure of efficacy of budesonide or dexamethasone.
The numbers of bronchoscopies | 2 days
  The bronchoscopy will demonstrate the non-inflammatory causes of stridor, such as: vocal cord paralysis, granuloma formation, subglottic stenosis, cricoarytenoid joint disfunction. In these cases, neither dexamethasone nor budesonide will improve clinical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela NM Medeiros, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Instituto Israelita de Ensino e Pesquisa Albert Einstein 's (IIEP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Klassen TP, Feldman ME, Watters LK, Sutcliffe T, Rowe PC. Nebulized budesonide for children with mild-to-moderate croup. N Engl J Med. 1994 Aug 4;331(5):285-9. doi: 10.1056/NEJM199408043310501. PMID 8022437
- [Background] Johnson DW, Jacobson S, Edney PC, Hadfield P, Mundy ME, Schuh S. A comparison of nebulized budesonide, intramuscular dexamethasone, and placebo for moderately severe croup. N Engl J Med. 1998 Aug 20;339(8):498-503. doi: 10.1056/NEJM199808203390802. PMID 9709042
- [Background] Geelhoed GC, Macdonald WB. Oral and inhaled steroids in croup: a randomized, placebo-controlled trial. Pediatr Pulmonol. 1995 Dec;20(6):355-61. doi: 10.1002/ppul.1950200604. PMID 8649914
- [Background] Sinha A, Jayashree M, Singhi S. Aerosolized L-epinephrine vs budesonide for post extubation stridor: a randomized controlled trial. Indian Pediatr. 2010 Apr;47(4):317-22. doi: 10.1007/s13312-010-0060-z. Epub 2009 Sep 3. PMID 19736368